CLINICAL TRIAL: NCT01218594
Title: Phase I/II Clinical Trial of Recombinant Human Endostatin in Combination With Concurrent Chemo-Radiotherapy in the Patients With Unresectable Stage III Non-small-Cell Lung Cancer
Brief Title: Curative Effect Study of Endostatin Combined With Chemoradiotherapy to Non-small-cell Lung Cancer
Acronym: DP-EN-RT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other); Fujian Province Tumor Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); The Affiliated Tumor Hospital of Guangxi Medical University (Unknown); Zhejiang Cancer Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); The 458 Hospital of Chinese PLA (Other)
Responsible Party: Principal Investigator, Ming Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP-EN-RT
Record Dates: First submitted 2010-06-01; First posted 2010-10-11 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage III; Unresectable; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endostatin combine CCRT (Experimental): 7.5mg/m2,iv gtt daily up to 7 days,beginning 1 week before radiotherapy,and repeat every 2 weeks
  Interventions: Drug: Endostatin

INTERVENTIONS:
Drug: Endostatin — 7.5mg/m2,iv gtt daily up to 7 days,beginning 1 week before radiotherapy,and repeat every 2 weeks
  Other Names: Endostar

SUMMARY:
To evaluate the efficacy and safety of Endostar combined with concurrent chemo-radiotherapy (CCRT) in patients with unresectable stage III non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:To assess the treatment response rate (RR) of Endostar in combination with CCRT

Secondary

* The progression-free survival (PFS)
* The overall survival(OS).
* The failed treatment modality.
* The toxicity of this regimen.

OUTLINE CCRT:Patients receive chemotherapy comprising Docetaxel(65mg/m2,iv gtt duration>1h) and Cisplatin(65mg/m2,concurrent hydration) on days 1 and 29 and at least 3 hours after chemotherapy undergo concurrent 3D-CRT five days a week for total dose 60-66Gy.

Endostatin:Patients receive Endostatin 7.5mg/m2 daily by iv gtt up to 7 days consecutively 1 week before radiotherapy and repeat every 2 weeks.

Patients are seen in follow-up every 3 months for 2 years and then every 6 months thereafter. Physical examination and CT scans of the thorax and upper abdomen are performed routinely.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * untreated pathologically confirmed inoperable stage IIIA or IIIB NSCLC
  * weight loss of less than 10% in the past 6 months
  * performance status (PS) of 0 to 1
  * forced vital capacity in 1 second (FEV1) higher than 0.8 L
  * measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
  * absolute neutrophil count (ANC) of ≥ 1500/μL
  * hemoglobin ≥ 10 mg/dL
  * platelet ≥ 100,000/μL
  * serum creatinine ≤ 1.25 times of upper limit of normal (ULN)
  * calculated creatinine clearance (CrCl) of ≥ 60 ml/min
  * bilirubin 1.5×ULN
  * AST and ALT less than 2.5×ULN
  * alkaline phosphatase less than 5×ULN.

Exclusion Criteria:

* active infection
* history of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* malnutrition (loss of ≥ 20% of the original body weight)
* sensor or motor neuropathy > grade I
* second primary malignancy, except for non-melanoma skin cancer
* psychiatric illness or social situation that would preclude study compliance
* pregnant or lactating women
* preexisting bleeding diatheses or coagulopathy
* Prior chemotherapy,chest irradiation therapy, or therapy directed at the epidermal growth factor receptor pathway

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, Doctor, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Bao Y, Peng F, Zhou QC, Yu ZH, Li JC, Cheng ZB, Chen L, Hu X, Chen YY, Wang J, Wang Y, Ma HL, Xu ZM, Lu RB, Deng XW, Chen M. Phase II trial of recombinant human endostatin in combination with concurrent chemoradiotherapy in patients with stage III non-small-cell lung cancer. Radiother Oncol. 2015 Feb;114(2):161-6. doi: 10.1016/j.radonc.2014.11.039. Epub 2014 Dec 9. PMID 25497558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2009 and January 2012, 50 patients from 5 centers were enrolled onto the study.
Pre-assignment Details: Two patients refused treatment after consenting for therapy and were ultimately excluded from the trial before any treatment.
Groups:
- Endostar Plus CCRT: Patients received Endostar (7.5 mg/m2/d) through 7 days at weeks 1, 3, 5, and 7, and two cycles of docetaxel (65 mg/m2) and cisplatin (65 mg/m2) on days 8 and 36, with concurrent thoracic radiation at 60~66 Gy.
Period: Overall Study
Arm/Group | Endostar Plus CCRT
Started | 48
Completed | 36
Not Completed | 12
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Endostar Plus CCRT
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 38
Region of Enrollment [Number; unit: participants]
  China | 48

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Tumor response was evaluated with thoracic CT scans when CCRT was completed, in accordance with Response Evaluation Criteria in Solid Tumors Group (RECIST).
Time Frame: 4 weeks after CCRT
Population: Response rate (RR)include complete response and partial response.
Measure: Number; unit: percentage of participants
Arm/Group | Endostar Plus CCRT
Number analyzed (Participants) | 48
percentage of participants | 37

ADVERSE EVENTS:
Arm/Group | Endostar Plus CCRT
Serious Adverse Events (participants affected / at risk) | 2/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endostar Plus CCRT (N=48)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
special pneumohemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endostar Plus CCRT (N=48)
Hematologic toxicity (Blood and lymphatic system disorders) | 47 (47)
Dermatology (Skin and subcutaneous tissue disorders) | 47 (47)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 43 (43)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20 (20)
Vomiting (Gastrointestinal disorders) | 19 (19)

LIMITATIONS AND CAVEATS:
This was a single-arm study, no comparison between Endostar to CCRT and CCRT alone was performed. It is not clear whether the observed improvement in survival is a result of the addition of Endostar or patient selection.The patient samples are small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No